CLINICAL TRIAL: NCT00865150
Title: How Illness and Nutritional Support Influence Amino Acid and Acylcarnitine Profiles in Premature Neonates
Brief Title: Amino Acid and Acylcarnitine Profiles in Premature Neonates
Status: Completed | Type: Observational
Sponsor: Pediatrix (Other)
Responsible Party: Sponsor
Other Study IDs: PDX-001-08
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Last update posted 2012-03-01 (Estimated); Status verified 2012-02

CONDITIONS: Prematurity; Neonatal Screening; Parenteral Nutrition
Keywords: Prematurity; Neonatal screening; Parenteral nutrition; Amino acids; Acylcarnitine
MeSH Terms: conditions — Premature Birth; Hyperphagia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Primary Hypotheses of the study include:

* Metabolic profiles are influenced by gestational age, chronological age, type and degree of nutritional support and illness
* Metabolic profiles differ between neonates who receive commercial formula and neonates who receive primarily human breast milk
* Neonates who develop parenteral associated cholestasis have metabolic markers that identify at risk patients (high serum urea nitrogen, citrulline, histidine, methionine, and succinyl carnitine and low thyroxine, serine and glutamate)
* Neonates that have hypothyroidism have abnormal metabolic profiles (low tyrosine levels)

DETAILED DESCRIPTION:
Malnutrition is a common problem in the neonatal intensive care unit. Recent studies indicate that prematurely born neonates commonly develop a severe nutritional deficit during the first weeks after birth, referred to as extrauterine growth restriction. Despite an increase in growth during the second month of hospitalization, many neonates are ultimately discharged home having grown inadequately. The early nutritional deficit affects weight gain as well as growth in length and head circumference. Aggressive administration of parenteral amino acids to improve protein accretion rates in very preterm neonates has been supported in the literature. Although tolerance of high dose amino acids has been described, researchers acknowledge that sensitive tests to monitor amino acid toxicity are not readily available in the clinical setting.

The goals of this study are:

* To better define normal amino acid and acylcarnitine values and how they change in premature neonates
* To measure the effect nutritional support has (human breastmilk vs. formula) on amino acid and acylcarnitines profiles
* To measure the effect of illness (parenteral nutrition associated cholestasis) on amino acid and acylcarnitine profiles
* To better define abnormal metabolic profiles (low tyrosine levels) in neonates that have hypothyroidism.

ELIGIBILITY:
Inclusion Criteria

* Documentation of informed consent
* Inborn
* Less than or equal to twenty four (24) hours of age
* Gestational age between twenty three (23) weeks and 0/7 days and thirty one (31) weeks and 0/7 days as per the best estimate by the neonatologist
* If subject is transferred to another hospital, the ability to obtain follow-up data on outcomes
* No known major anomalies (inborn error of metabolism, chromosomal abnormalities, cyanotic congenital heart disease, gastroschisis, omphalocele, diaphragmatic hernia or other major gastrointestinal anomalies, major neurological injury or anomaly, and multiple congenital anomalies)

Exclusion Criteria

* Outborn (transferred for intensive care from another hospital)
* Greater than twenty four (24) hours of age
* Gestational age < 23 weeks or > 31 weeks
* Any known major congenital anomalies

Ages: 23 Weeks to 31 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Hospital
Sampling Method: Probability Sample
Enrollment: 1003 (Actual)
Dates: Start 2009-04; Primary Completion 2011-08 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Metabolic Profile - Serum amino acid, acylcarnitine and thyroxine levels. Day of birth, (first 24 hours), Day 7, (parenteral nutrition effect), Day 28, (enteral nutrition effect), Day 42, or discharge (established enteral feeding and growth) | 42 Days of Life

SECONDARY OUTCOMES:
Occurrence of any of the following: death, cholestatic liver disease, positive blood or CSF culture, NEC, IVH, or respiratory support at 36 weeks PMA. | 42 Days of Life

CONTACTS AND LOCATIONS:
Overall Officials: Reese Clark, MD, Principal Investigator — Pediatrix Medical Group, Inc.
Locations (2):
- United States (2):
  - Memorial Hospital South Bend, South Bend, Indiana
  - McLeod Regional Medical Center, Florence, South Carolina

REFERENCES:
- [Derived] Clark RH, Chace DH, Spitzer AR. Impact of l-carnitine supplementation on metabolic profiles in premature infants. J Perinatol. 2017 May;37(5):566-571. doi: 10.1038/jp.2016.253. Epub 2017 Jan 12. PMID 28079870
- [Derived] Jacob J, Kamitsuka M, Clark RH, Kelleher AS, Spitzer AR. Etiologies of NICU deaths. Pediatrics. 2015 Jan;135(1):e59-65. doi: 10.1542/peds.2014-2967. Epub 2014 Dec 8. PMID 25489010